CLINICAL TRIAL: NCT01372852
Title: Plasma Adiponectin Concentration, Activity and Isoforms in Newly Diagnosed and Untreated T2DM Patients in Chinese Population
Brief Title: Plasma Adiponectin Concentration, Activity and Isoforms in Newly Diagnosed and Untreated Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Ling Tao, Department of Cardiology of Xijing Hospital; Fourth Military Medical University
Other Study IDs: xjyy110501
Record Dates: First submitted 2011-06-11; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood，abdominal fat tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2DM patients: newly diagnosed T2DM patients and untreated with any drugs.
- Non-diabetic Control Group

SUMMARY:
The objective of present study were to compare plasma adiponectin isoform status, their bioactivities newly diagnosed Chinese with healthy volunteer.

DETAILED DESCRIPTION:
Adiponectin, circulates as trimer, hexamer and high molecular weight form (HMW) in human blood, is a promising biomarker for indication diabetes and cardiovascular disease. Both adiponectin complexes concentration and their bioactivities are decreased in pathological state. Disulﬁde-bond A oxidoreductase-like protein (DsbA-L) is a key regulator for adiponectin biosynthesis and its expression level is down-regulated in obese mice and humans. However, the alteration of circulating adiponectin multimers distribution, their bioactivities and adiponectin regulator, DsbA-L level, in newly diagnosed Chinese type 2 diabetes patients are unknown. The objective of present study were to compare plasma adiponectin isoform status, their bioactivities and DsbA-L concentration in newly diagnosed Chinese with healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Having a diabetic history within 12 months
* BMI smaller than 30kg/m2

Exclusion Criteria:

* Having any kinds of treatment affecting glucose
* pregnant
* uncontrolled hypertension, active cardiac disease, or other major liver, kidney disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls a group of 30-70years patients from primary care clinic who have diabetes history within 12 months and without taking any treatment.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
plasma adiponectin concentration, isoform distribution and activity. | participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D Ph.D, Principal Investigator — Department of Cardiology of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China